CLINICAL TRIAL: NCT00001011
Title: The Safety and Efficacy of Zidovudine in the Treatment of Patients With Early AIDS Related Complex
Brief Title: The Safety and Effectiveness of Zidovudine in the Treatment of Patients With Early AIDS Related Complex
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 016; 10992 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Virus Replication; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To determine the safety and usefulness of zidovudine (AZT) for the treatment of patients with early symptomatic HIV infection or early AIDS related complex (ARC). The ability of AZT to suppress HIV, to improve body defenses, and to prevent the occurrence or development of AIDS or advanced ARC is being evaluated.

In one human study, patients with AIDS or advanced ARC who received AZT had fewer life-threatening infections, improved in weight and performance, and lived longer than patients who received a placebo (inactive medication). Further studies are needed because toxic effects associated with the use of AZT were noted and the long-term effectiveness and toxicity of AZT are still unknown. It is also unknown if AZT will benefit patients with less severe HIV infections such as early ARC or PGL.

DETAILED DESCRIPTION:
In one human study, patients with AIDS or advanced ARC who received AZT had fewer life-threatening infections, improved in weight and performance, and lived longer than patients who received a placebo (inactive medication). Further studies are needed because toxic effects associated with the use of AZT were noted and the long-term effectiveness and toxicity of AZT are still unknown. It is also unknown if AZT will benefit patients with less severe HIV infections such as early ARC or PGL.

Patients accepted into the study are randomly assigned to receive either AZT or placebo. Treatment continues for a minimum of 104 weeks beyond the time the last patient enters the study. If the study medication causes toxic effects, the dose is decreased or temporarily stopped, and if the toxic effects are severe, then the medication will be stopped permanently. Participants visit the clinic every 2 weeks during the first 16 weeks and once a month thereafter. Throughout the study frequent blood samples are taken to monitor the effectiveness and safety of the treatment. AMENDED: The placebo arm has been discontinued as of August 3, 1989 and the AZT dose has been reduced.

ELIGIBILITY:
Inclusion Criteria

* Patients must have a positive antibody to HIV confirmed by a federally licensed ELISA test kit.
* The CD4 cell count must be 201 - 799 cells/mm3 measured on two separate occasions within 60 days at least 72 hours apart prior to study entry (at least 1 of 2 counts and the mean must be < 800 cells/mm3, and at least 1 of 2 counts and the mean must be > 200 cells/mm3). The last count must be within 14 days of study entry.

Concurrent Medication:

Allowed:

* Acetaminophen and acetaminophen products but use should be minimized. Continuous use for > 72 hours is discouraged.
* Aerosolized pentamidine.

Prior Medication:

Allowed:

* Chemoprophylaxis for Pneumocystis carinii pneumonia with aerosolized pentamidine of 300 mg every 4 weeks through the Respirgard II nebulizer if patient has CD4(+) count < 200 cells/mm3 measured on 2 determinations at least 48 hours apart.

Exclusion Criteria

Concurrent Medication:

Excluded:

* Other antiretroviral agents, biologic modifiers or corticosteroids.
* Other experimental medications.
* Systemic chemoprophylaxis of Pneumocystic carinii pneumonia (PCP) - aerosolized pentamidine is allowed.

Prior Medication:

Excluded:

* Zidovudine (AZT).
* Other antiretroviral agents.
* Excluded within 30 days of study entry:
* Biologic modifiers or corticosteroids.
* Excluded within 60 days of study entry:
* Ribavirin.

Prior Treatment:

Excluded within 30 days of study entry:

* Blood transfusions.

Patients may not have any of the following diseases or symptoms:

* Active oral candidiasis at entry.
* An opportunistic infection or malignancy fulfilling the definition of AIDS (CDC Surveillance Case Definition for Acquired Immunodeficiency Syndrome).
* Temperature > 38.5 degrees C persisting for > 14 consecutive days or > 15 days in a 30-day interval present at entry.
* Chronic diarrhea defined as = or > 3 liquid stools per day, persisting for > 14 days without a definable cause during the past 2 years.
* HIV neurologic disease as manifested by motor abnormalities including impaired rapid eye movements or ataxia; motor weakness in the lower extremities; sensory deficit consistent with a peripheral neuropathy; bladder or bowel incontinence.
* Concurrent neoplasms other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Subjects with hemophilia should be evaluated and treated under the hemophilia protocols, if available at that ACTG.

Patients may not have any of the following diseases or symptoms:

* Active oral candidiasis at entry.
* An opportunistic infection or malignancy fulfilling the definition of AIDS (CDC Surveillance Case Definition for Acquired Immunodeficiency Syndrome).
* Temperature > 38.5 degrees C persisting for > 14 consecutive days or > 15 days in a 30-day interval present at entry.
* Chronic diarrhea defined as = or > 3 liquid stools per day, persisting for > 14 days without a definable cause during the past 2 years.
* HIV neurologic disease as manifested by motor abnormalities including impaired rapid eye movements or ataxia; motor weakness in the lower extremities; sensory deficit consistent with a peripheral neuropathy; bladder or bowel incontinence.
* Concurrent neoplasms other than basal cell carcinoma of the skin or in situ carcinoma of the cervix.
* Subjects with hemophilia should be evaluated and treated under the hemophilia protocols, if available at that ACTG.

Active drug or alcohol abuse.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 538
Dates: Study Completion 1995-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MA Fischl, Study Chair; DD Richman, Study Chair
Locations (40):
- United States (40):
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Harbor UCLA Med Ctr, Torrance, California
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - St Louis Regional Hosp / St Louis Regional Med Ctr, St Louis, Missouri
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Columbus Children's Hosp, Columbus, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Fischl MA, Richman DD, Hansen N, Collier AC, Carey JT, Para MF, Hardy WD, Dolin R, Powderly WG, Allan JD, et al. The safety and efficacy of zidovudine (AZT) in the treatment of subjects with mildly symptomatic human immunodeficiency virus type 1 (HIV) infection. A double-blind, placebo-controlled trial. The AIDS Clinical Trials Group. Ann Intern Med. 1990 May 15;112(10):727-37. doi: 10.7326/0003-4819-112-10-727. PMID 1970466
- [Background] Bass HZ, Hardy WD, Mitsuyasu RT, Wang YX, Cumberland W, Fahey JL. Eleven lymphoid phenotypic markers in HIV infection: selective changes induced by zidovudine treatment. J Acquir Immune Defic Syndr (1988). 1992;5(9):890-7. PMID 1512689
- [Background] Bass HZ, Nishanian P, Hardy WD, Mitsuyasu RT, Esmail E, Cumberland W, Fahey JL. Immune changes in HIV-1 infection: significant correlations and differences in serum markers and lymphoid phenotypic antigens. Clin Immunol Immunopathol. 1992 Jul;64(1):63-70. doi: 10.1016/0090-1229(92)90060-2. PMID 1376654
- [Background] Wu AW, Rubin HR, Mathews WC, Brysk LM, Bozzette SA, Hardy WD, Atkinson JH, Grant I, Spector SA, McCutchan JA, et al. Functional status and well-being in a placebo-controlled trial of zidovudine in early symptomatic HIV infection. J Acquir Immune Defic Syndr (1988). 1993 May;6(5):452-8. PMID 8483109
- [Background] Jacobson MA, Gundacker H, Hughes M, Fischl M, Volberding P. Zidovudine side effects as reported by black, Hispanic, and white/non-Hispanic patients with early HIV disease: combined analysis of two multicenter placebo-controlled trials. J Acquir Immune Defic Syndr Hum Retrovirol. 1996 Jan 1;11(1):45-52. doi: 10.1097/00042560-199601010-00006. PMID 8528732
- [Background] Kozal MJ, Shafer RW, Winters MA, Katzenstein DA, Merigan TC. A mutation in human immunodeficiency virus reverse transcriptase and decline in CD4 lymphocyte numbers in long-term zidovudine recipients. J Infect Dis. 1993 Mar;167(3):526-32. doi: 10.1093/infdis/167.3.526. PMID 7680058
- [Background] McCorkindale C, Dybevik K, Coulston AM, Sucher KP. Nutritional status of HIV-infected patients during the early disease stages. J Am Diet Assoc. 1990 Sep;90(9):1236-41. PMID 2168908
- [Background] Lin DY, Fischl MA, Schoenfeld DA. Evaluating the role of CD4-lymphocyte counts as surrogate endpoints in human immunodeficiency virus clinical trials. Stat Med. 1993 May 15;12(9):835-42. doi: 10.1002/sim.4780120904. PMID 8101011
- [Background] Lagakos S, Fischl MA, Stein DS, Lim L, Volberding P. Effects of zidovudine therapy in minority and other subpopulations with early HIV infection. JAMA. 1991 Nov 20;266(19):2709-12. PMID 1942422
- [Background] Melnick SL, Hannan P, Decher L, Little JW, Rhame FS, Balfour HH Jr, Volberding P. Increasing CD8+ T lymphocytes predict subsequent development of intraoral lesions among individuals in the early stages of infection by the human immunodeficiency virus. J Acquir Immune Defic Syndr (1988). 1991;4(12):1199-207. PMID 1682473